CLINICAL TRIAL: NCT05274191
Title: An Exploratory Basket Study of Pyrotinib Maleate Tablets in HER2 Mutated or Amplified of Metastatic Solid Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhongshan Hospital Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-228
Record Dates: First submitted 2022-03-02; First posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Solid Tumor
Keywords: HER2 mutation or amplification,Pyrotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A single arm, open-label Phase II clinical study. (Experimental): All subjects enrolled will receive the following treatment：Pyrotinib±standard treatment.
  Pyrotinib 400 mg/ D (once a day, at the same time each day) until the progression of disease; Chemotherapy regimens follow the programme cycle recommended by the guidelines or as determined by the investigator.
  The dosage can be adjusted according to the protocol according to the adverse reactions of subjects. Subjects will continue to take medication until completion of the prescribed course of treatment, disease progression, toxicity intolerance, withdrawal of Informed Consent Form, or termination in the investigator's judgment.
  Interventions: Drug: Pyrotinib Maleate; Other: standard regimen

INTERVENTIONS:
Drug: Pyrotinib Maleate — Pyrotinib ± standard regimen Pyrotinib: 400 mg/day (once a day, orally at the same time every day), continued until disease progression;
Other: standard regimen — standard regimen

SUMMARY:
A single arm, open-label Phase II clinical study.The subjects were patients with lung, gastric and colorectal cancers.

DETAILED DESCRIPTION:
Object: 1.The main purpose: T To observe and evaluate the efficacy of pyrotinib in patients with HER2-mutated/amplified metastatic solid tumors after failure of standard therapy; 2. Secondary objectives: To observe and evaluate the safety of pyrotinib in patients in HER2 mutated or amplified metastatic solid tumors after failure of standard treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18-75 years old, regardless of gender;
2. Disease progression during the previous standard treatment or disease progression within 6 months after the end of treatment, patients with gastric and gastroesophageal junction adenocarcinoma requires previous use of trastuzumab, and other tumors must have received at least first-line standard chemotherapy ± targeted therapy.
3. Two or more grade IV hematological toxicity or non-hematological toxicity ≥ grade III or damage to the heart, liver, kidney and other major organs of grade ≥ II occurred during the standard treatment process; Patients who have been confirmed by the doctor to no longer receive standard treatment can be included in the group.
4. HER2 mutated non-small cell lung cancer , gastric and gastroesophageal junction adenocarcinoma or Adenocarcinoma of the colon has been confirmed by Pathology.
5. Cancer tissue pathology is clearly HER2 positive: including IHC2+/ISH+, IHC 3+ or HER2 mutations (the results obtained by NGS method, PCR method, Sanger method, mass spectrometry sequencing and other measurement methods are all acceptable).
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
7. For recurrent or metastatic tumours, according to the RECIST 1.1 standard, the subject has at least one measurable target disease.
8. Life expectancy greater than or equal to 12 months;
9. The functional level of organs must meet the following requirements:

(1) Blood routine: ANC ≥ 1.5×10^9/L; PLT ≥ 90×10^9/L; Hb ≥ 90 g/L; (2) Blood biochemistry: TBIL<=1.5×ULN; ALT and AST<=2×ULN; for subjects with liver metastases, ALT and AST<=5×ULN; BUN and Cr<=1.5×ULN and creatinine clearance ≥50mL/min (Cockcroft-Gault formula); (3) Heart color Doppler ultrasound: LVEF≥50%; (4) 12-lead electrocardiogram: The QT interval (QTcF) corrected by Fridericia's method is <450ms for males and <470ms for females.

10. Have sufficient bone marrow, liver and kidney functions. 11. Women of childbearing age and their spouses are willing to contraception during treatment and within 1 year after the last medication.

Volunteer to join the study, sign an informed consent form, have good compliance and are willing to cooperate with follow-up.

Exclusion Criteria:

* 1. Left ventricular ejection fraction (LVEF) < 50% at baseline (measured by echocardiography or MUGA); 2. Patients who have received systemic therapy including immunotherapy, biotherapy and any clinical trial drugs in the past 2 weeks; 3. Patients with uncontrollable central metastases, brain tumor lesions confirmed by brain CT or MRI and need dehydration treatment or radiotherapy (except for patients with stable brain metastases after 1 month of radiotherapy); 4. With > grade 1 unresolved toxicity due to any previous treatment / procedure (ctc-ae, except alopecia, anemia, and hypothyroidism); 5. Severe infection and other serious systemic diseases; 6. Patients receiving long-term or high-dose corticosteroid treatment (inhaled steroids or short-term oral steroids are allowed to resist vomiting or promote appetite); 7. Evidence or history of coagulation disorders such as bleeding events with grade ≥ 3 (ctc-ae); 8. Patients whom intestinal obstruction and other factors affecting oral administration or absorption of drugs; After the comprehensive judgment of the disease, the researcher thought that it was not suitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-04 (Estimated); Primary Completion 2022-03-15 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 24 months
  Defined as proportion of complete response and partial response according to RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Overall survival | 24 months
  Defined as the time from the date of informed consent until to the date of death, regardless of the cause of death.
Disease control rate | 24 months
  the proportion of patients whose tumors shrink or remain stable for a certain period of time, including complete remission (CR), partial remission (PR) and stable (SD) cases
Progression-free survival | 24 months
  Defined as the time from the date of informed consent to first documented disease progression (PD) using Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) or death from any cause, whichever occurred first.

CONTACTS AND LOCATIONS:
Overall Officials: li xiao, Principal Investigator — Zhongshan Hospital Affiliated to Xiamen University